CLINICAL TRIAL: NCT02186223
Title: The Angel® Catheter Clinical Trial: Prevention of Pulmonary Embolism in High Risk Subjects
Brief Title: The Angel® Catheter Pivotal Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BiO2 Medical (Industry)
Collaborators: CardioMed Device Consultants, LLC (Industry); Intrinsic Imaging, LLC (Unknown); Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QD-230
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboembolism; Trauma
Keywords: Pulmonary Embolism; PE; DVT; Deep Vein Thrombosis; VTE; Venous Thromboembolism; prophylaxis; thromboprophylaxis; contraindications to thromboprophylaxis; prophylactic; prevention; Inferior vena cava filter; IVC filter; filter; prevention of pulmonary embolism; trauma; critically-ill
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism; Wounds and Injuries; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The Angel® Catheter (Experimental): All eligible subjects will receive an Angel® Catheter.
  Interventions: Device: The Angel® Catheter

INTERVENTIONS:
Device: The Angel® Catheter — The Angel® Catheter is a temporary device that combines the functions of an inferior vena cava (IVC) filter and a 3-lumen central venous catheter (CVC). The device can be placed at the bedside into the inferior vena cava via the femoral vein for the prevention of Pulmonary Embolism (PE) and for access to the central venous system. The device is intended for short-term (less than 30 days) vascular access via the femoral vein.

SUMMARY:
The primary objective of this multicenter, prospective, single arm clinical trial is to evaluate the safety and effectiveness of the Angel® Catheter in subjects at high risk of PE, and with recognized contraindications to standard pharmacological therapy (anticoagulation).

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative is willing and able to provide written informed consent,
2. Subject is 18 years or older,
3. Subject is expected to remain in a critical care setting for at least 72 hours,

   AND at least one of the following inclusion criteria (4,5, and/or 6)
4. Subject has recognized contraindications to standard pharmacological thromboprophylaxis including:

   * Active bleeding or at high risk for bleeding OR
   * Hypersensitivity to pharmacological thromboprophylaxis OR
   * History of severe heparin induced thrombocytopenia OR
   * Severe thrombocytopenia
5. Subject has a confirmed acute proximal lower extremities DVT or a confirmed acute PE with recognized contraindication to anticoagulation
6. Subject requires a temporary interruption (>24 hours) of pharmacological thromboprophylaxis for a surgical or medical procedure

Exclusion Criteria:

1. Subject is pregnant
2. Subject is in treatment with an investigational drug or device within 30 days prior to enrollment
3. Subject has a pre-existing IVC filter in place
4. BMI = > 45
5. Subject has functioning pelvic renal allograft on the only side available for device insertion
6. Subject has undergone a surgical procedure involving the femoral vein or pelvic veins through which the device must be inserted
7. Anatomic inability to place the Angel® Catheter
8. Subject has known hypersensitivity to any of the components of the Angel® Catheter, specifically Nitinol (nickel and/or titanium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tapson, MD, Principal Investigator — Cedars Sinai
Locations (21):
- United States (21):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC San Diego Medical Center, San Diego, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Delray Medical Center, Delray Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - University of New Mexico Health, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Regional One Health, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - John Peter Smith Health Network, Fort Worth, Texas
  - Ben Taub Hospital, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Angel® Catheter
Started ((i.e., consented)) | 172
Device Placed | 163
Completed ((i.e., Device in place for at least 48 hours)) | 151
Not Completed | 21
Not completed — Not eligible for device placement | 6
Not completed — Unable to obtain femoral access | 3
Not completed — Death | 3
Not completed — Device in place less than 48 hours | 9

BASELINE CHARACTERISTICS:
Population: Population includes all subjects that had the Angel® Catheter placed.
Groups:
- The Angel® Catheter: All eligible subjects received an Angel® Catheter.
  The Angel® Catheter: The Angel® Catheter is a temporary device that combines the functions of an inferior vena cava (IVC) filter and a 3-lumen central venous catheter (CVC). The device can be placed at the bedside into the inferior vena cava via the femoral vein for the prevention of Pulmonary Embolism (PE) and for access to the central venous system. The device is intended for short-term (less than 30 days) vascular access via the femoral vein.
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 139
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.07 (18.66)
Age, Customized [Median (Full Range); unit: years] | 43 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 122
  More than one race | 5
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 163
Time from admission to the hospital to admission to ICU [Mean (Standard Deviation); unit: hours] | 7.49 (27.34)
Time from admission to the hospital to admission to ICU [Median (Full Range); unit: hours] | 2.07 [0 to 292.33]
Primary ICU Admission Diagnosis [Count of Participants; unit: Participants]
  Trauma | 151
  Surgical | 2
  Medical | 6
  Neurological | 4
Type of trauma (for trauma subjects) [Count of Participants; unit: Participants] — Population: Number analyzed includes all trauma subjects that had an Angel® Catheter placed
  Participants
    Head/Spinal Trauma: number analyzed (Participants) | 151
    Head/Spinal Trauma | 129
    Chest: number analyzed (Participants) | 151
    Chest | 63
    Abdomen: number analyzed (Participants) | 151
    Abdomen | 41
    Lower Extremity Trauma: number analyzed (Participants) | 151
    Lower Extremity Trauma | 54
    More than one area affected: number analyzed (Participants) | 151
    More than one area affected | 80
    Head Bleed (Subcategory of Head/Spinal Trauma): number analyzed (Participants) | 129
    Head Bleed (Subcategory of Head/Spinal Trauma) | 102
Injury Severity Score (for trauma subjects) [Mean (Standard Deviation); unit: Injury Severity Score] — Injury Severity Score (ISS) Scale: Minimal (1-9); Moderate (10-15); Severe (16-24); Critical (25+); Trauma subjects categorized by their ISS, with higher scores representing more serious/life-threating injuries. This anatomical scoring system providing an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score and allocated to 1/6 body regions (Head, Face, Chest, Abdomen, Extremities & Pelvis, External). Highest score in each body region is used. 3 most severely injured regions have score squared and added to produce the ISS score. Population: Measure Analysis is specific only to trauma subjects.
  Injury Severity Score
    number analyzed (Participants) | 151
    (all) | 27.68 (11.94)
Injury Severity Score (for trauma subjects) [Median (Full Range); unit: Injury Severity Score] — Population: Number analyzed includes all trauma subjects that had an Angel® Catheter placed
  Injury Severity Score
    number analyzed (Participants) | 151
    (all) | 26 [5 to 66]
Injury Classification [Count of Participants; unit: Participants] — Trauma subjects were categorized based on their Injury Severity Score (ISS), with higher scores representing more serious or life-threating injuries. The ISS is an anatomical scoring system that provides an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score and allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities (including Pelvis), External). The highest AIS score in each body region is used. The 3 most severely injured body regions have their score squared and added together to produce the ISS score. Population: Number analyzed includes all trauma subjects that had the Angel® Catheter placed.
  Participants
    Minimal (1-9): number analyzed (Participants) | 151
    Minimal (1-9) | 7
    Moderate (10-15): number analyzed (Participants) | 151
    Moderate (10-15) | 11
    Severe (16-24): number analyzed (Participants) | 151
    Severe (16-24) | 41
    Critical (25+): number analyzed (Participants) | 151
    Critical (25+) | 92
Bleeding Risk [Count of Participants; unit: Participants]
  Active bleeding | 67
  History of bleeding | 13
  At high risk for bleeding | 69
Severity of Active Bleeding [Count of Participants; unit: Participants] — Population: Number analyzed includes all subjects with active bleeding at enrollment and subsequently had an Angel® Catheter placed.
  Participants
    Minor bleeding: number analyzed (Participants) | 67
    Minor bleeding | 11
    Major bleeding | 56
Medical History & Concomitant Conditions [Count of Participants; unit: Participants]
  Blood and lymphatic system disorders | 53
  Cardiac disorders | 43
  Endocrine disorders | 7
  Ear and labyrinth disorders | 2
  Eye disorders | 2
  Gastrointestinal disorders | 38
  General disorders and administration site conditio | 37
  Hepatobiliary disorders | 8
  Immune system disorders | 2
  Infections and infestations | 28
  Injury, poisoning, and procedural complications | 149
  Investigations | 43
  Metabolism and nutrition disorders | 58
  Musculoskeletal and connective tissue disorders | 26
  Neoplasms benign, malignant, and unspecified | 12
  Nervous system disorders | 111
  Psychiatric disorders | 24
  Renal and urinary disorders | 19
  Reproductive system and breast disorders | 11
  Respiratory, thoracic and mediastinal disorders | 101
  Skin and subcutaneous tissue disorders | 5
  Social circumstances | 3
  Surgical and medical procedures | 78
  Vascular disorders | 73
Subjects with Baseline Venous Thromboembolic (VTE) Disease per Site-reported Medical History [Count of Participants; unit: Participants]
  Pulmonary Embolism (PE) | 3
  Deep Vein Thrombosis (DVT) | 16
  PE and DVT | 1
Use of mechanical DVT preventive devices [Count of Participants; unit: Participants]
  At least 1 type of preventive device used | 145
  Compressive stockings | 10
  Pneumatic compression | 113
  Other | 27
Supplemental Oxygen at Enrollment [Count of Participants; unit: Participants] | 150
Type of supplemental oxygen [Count of Participants; unit: Participants] — Population: Number analyzed includes all patient receiving supplemental oxygen at enrollment that subsequently had an Angel® Catheter placed.
  Participants
    Mechanical ventilation: number analyzed (Participants) | 150
    Mechanical ventilation | 127
    CPAP-BiPAP: number analyzed (Participants) | 150
    CPAP-BiPAP | 0
    Nasal cannula/face mask: number analyzed (Participants) | 150
    Nasal cannula/face mask | 20
    Other: number analyzed (Participants) | 150
    Other | 2
Need for vasopressors before Angel® Catheter insertion [Count of Participants; unit: Participants] | 40
Other Central Venous Catheter (CVC) in place prior to Angel® Catheter insertion [Count of Participants; unit: Participants]
  None | 46
  Short term CVC | 109
  Long term CVC | 8
Indications for the Angel® Catheter Placement [Count of Participants; unit: Participants]
  Recognized contraindications to anticoagulation | 160
  Acute LE DVT or PE & contraindicated to anticoagul | 8
  Temporary interruption of anticoagulation | 10
  Prophylactic Use of Indications for the Angel® Cat | 160
Contraindications to anticoagulation [Count of Participants; unit: Participants] — Population: Number analyzed includes all subjects that had recognized contraindications to standard pharmacological thromboprophylaxis reported.
  Participants
    Active or high risk for bleeding: number analyzed (Participants) | 160
    Active or high risk for bleeding | 153
    Hypersensitivity to anticoagulation: number analyzed (Participants) | 160
    Hypersensitivity to anticoagulation | 0
    History of severe heparin induced thrombocytopenia: number analyzed (Participants) | 160
    History of severe heparin induced thrombocytopenia | 0
    Severe thrombocytopenia: number analyzed (Participants) | 160
    Severe thrombocytopenia | 1
    Other: number analyzed (Participants) | 160
    Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Clinically Significant PE or Fatal PE During Treatment Period
Description: 1. Clinically Significant PE: Subjects will be assessed daily for signs and symptoms of PE. If present and no alternative diagnosis is suspected, at least one of four defined diagnostic examinations will performed to confirm or rule out PE.
  2. Fatal PE: Defined as unexpected death within 24 hours of onset of the acute event with a verified initial symptomatic DVT or PE where there is no other reasonable cause of death.
Time Frame: Assessed daily from Baseline through Study Exit which occurs 3 days post-Angel Catheter Removal OR at hospital discharge, whichever is first (maximum of 33 assessment days with an anticipated average of 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Participants | 163

2. Secondary Outcome: Incidence of Acute Proximal Deep Vein Thrombosis
Time Frame: Assessed daily from Baseline through Study Exit which occurs 3 days post-Angel Catheter Removal OR at hospital discharge, whichever occurs first (maximum of 33 assessment days with an anticipated average of 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Participants | 30

3. Secondary Outcome: Incidence of Catheter Related Thrombosis
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Participants | 20

4. Secondary Outcome: Incidence of Catheter Related Blood Stream Infections
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Participants | 0

5. Secondary Outcome: Incidence of Major Bleeding Event
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | The Angel® Catheter
Number analyzed (Participants) | 163
Participants | 5

6. Secondary Outcome: Incidence of PEs Averted
Description: During the pre-removal cavogram, the presence of significant clot (>25% of the volume of the filter) trapped by the Angel® Catheter will be assessed. The number of subjects with significant clot trapped by the device will be reported as the number of PEs averted.
Time Frame: During the pre-removal cavogram (An average of 6.8 days after device insertion)
Measure: Count of Participants; unit: Participants
Groups:
- Angel® Catheter Pre-Removal Cavogram: Number analyzed includes all subjects that had an Angel® Catheter placed, and a cavogram was performed prior to removal.
Arm/Group | Angel® Catheter Pre-Removal Cavogram
Number analyzed (Participants) | 129
Participants | 14

ADVERSE EVENTS:
Time Frame: From the time of Angel® Catheter insertion, through the entire catheter indwelling period (Mean±SD: 6.79±3.97 days; Median(Range: Min,Max): 5.94 (0.34,21.92) days), until death, discharge or 3 days post-removal, whichever occurs first.
Arm/Group | The Angel® Catheter
Serious Adverse Events (participants affected / at risk) | 49/163
Other Adverse Events (participants affected / at risk) | 114/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Angel® Catheter (N=163)
Cardiac Arrest (Cardiac disorders) | 4 (4)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Brain Death (General disorders) | 2 (2)
Multi-Organ Failure (General disorders) | 3 (3)
Chronic Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 4 (4)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Brain Hypoxia (Nervous system disorders) | 1 (1)
Brain Oedema (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Intracranial Pressure Increased (Nervous system disorders) | 5 (5)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Deep Vein Thrombosis (Vascular disorders) | 10 (10)
Haemodynamic Instability (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pelvic Venous Thrombosis (Vascular disorders) | 2 (2)
Vena Cava Thrombosis (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Angel® Catheter (N=163)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 2 (2)
Axillary vein thrombosis (Vascular disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 5 (5)
Bacterial vaginosis (Infections and infestations) | 2 (2)
Blood albumin decreased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 2 (2)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Catheter site haemorrhage (General disorders) | 1 (1)
Central nervous system infection (Infections and infestations) | 1 (1)
Cerebral hypoperfusion (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Clostridium test positive (Investigations) | 3 (3)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Culture urine positive (Investigations) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 15 (15)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Device damage (General disorders) | 1 (1)
Device deployment issue (General disorders) | 1 (1)
Device dislocation (General disorders) | 3 (3)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diffuse axonal injury (Injury, poisoning and procedural complications) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Gastric hypomotility (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (5)
Hyperthermia (General disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 9 (9)
Hypoxia (Vascular disorders) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 2 (2)
Klebsiella test positive (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lobar pneumonia (Infections and infestations) | 2 (2)
Local swelling (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (4)
Melaena (Gastrointestinal disorders) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myoglobinuria (Renal and urinary disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Platelet count increased (Vascular disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 24 (24)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia psudomonal (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulse absent (Investigations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scleral oedema (Eye disorders) | 1 (1)
Secondary hypertension (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 3 (3)
Tracheobronchitis (Infections and infestations) | 2 (2)
Unintentional medical device removal (General disorders) | 12 (12)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (9)
Vena cava thrombosis (Vascular disorders) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days